CLINICAL TRIAL: NCT00904085
Title: A Randomized, Double-blind Evaluation of the Analgesic Efficacy and Safety of a Low Dose Oxymorphone Immediate Release in Patients Following Ambulatory Arthroscopic Knee Surgery
Brief Title: Post-operative Efficacy and Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EN3203-008
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymorphone (Active Comparator)
  Interventions: Drug: Oxymorphone IR
- Placebo (Placebo Comparator)
  Interventions: Drug: Oxymorphone IR

INTERVENTIONS:
Drug: Oxymorphone IR — 5 mg

SUMMARY:
The purpose of this study was to compare the analgesic efficacy of 5 mg oxymorphone IR with placebo in patients with mild to moderate pain following outpatient knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years of age or older, who have completed outpatient knee arthroscopy
* Have an initial pain intensity score of between 30mm and 70mm on a 100mm Visual Analogue Scale(VAS) and a categorical pain rating scale of none, mild, moderate, or severe,
* Have been informed of the nature of the study and provided written informed consent

Exclusion Criteria:

* Have a positive pregnancy test
* Have received any of the following medications within 24 hours prior to dosing: COX2 inhibitors, Minor Tranquilizers, Muscle relaxants, Antihistamines
* Long-acting oral and parenteral analgesics are prohibited for at least 12 hours prior to receiving study medication.
* Have received any of the following medication within 48 hours prior to dosing: Chronic use of analgesics (opioid or non-opioid including aspirin [>325 mg/day], acetaminophen, and NSAIDs)
* Have received MAOI drugs within 2 weeks prior to dosing
* Not stabilized on the following medications for at least 4 weeks prior to dosing: Tricyclic antidepressant drugs, Serotonin reuptake inhibitors, Amphetamines used for ADHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2003-04; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity (SPID) Visual Analog Scale (VAS) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals